CLINICAL TRIAL: NCT03270306
Title: Eating Behaviours, Diet Quality and Gastrointestinal Symptoms in Children With Autism Spectrum Disorders and Typically Developing Children: a Case-control Study
Brief Title: Eating Behaviours, Diet and Gastrointestinal Symptoms in Children With Autism Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ruth Chan, Senior Research Fellow, Chinese University of Hong Kong
Other Study IDs: 2016.607
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Stool sample and blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This case-control study aims to compare the differences in eating behaviours, nutritional status, diet quality and gastrointestinal (GI) health between Chinese children aged 3-6 years with autism spectrum disorders (ASD) (n=65) and typically developing children (TDC) (n=65).

DETAILED DESCRIPTION:
Objective: To compare the differences in eating behaviours, nutritional status, diet quality and gastrointestinal (GI) health between Chinese children aged 3-6 years with autism spectrum disorders (ASD) and typically developing children (TDC).

Hypotheses:

1. Children with ASD will show more problematic mealtime behaviours as represented by higher scores of 'limited variety' and 'food refusal' domains of the BAMBI compared to typically developing children
2. Children with ASD will have more GI symptoms, in particular constipation and diarrhea compared to typically developing children
3. Children with ASD will have a lower ratio of Bacteroidetes to Firmicutes than the typical control children
4. Children with ASD will have less desirable diet quality in terms of lower dietary index, lower dietary diversity score and lower intake of fibre, iron, calcium, zinc and vitamin C compared to typically developing children
5. A better diet quality will be associated with a more favourable gut microbial composition in children with and without ASD

Design and subjects: Case-control study including 65 families with children of ASD and 65 families with TDC matched by child's age and sex.

Outcomes: The primary outcomes will be the difference in mean scores of 'limited variety' and 'food refusal' domains of the Chinese version of BAMBI between children with ASD and typically developing children. The secondary outcomes will be the difference in the occurrence of GI symptoms in terms of constipation and diarrhea, as well as the difference in the gut microbiota profile in terms of the Bacteroidetes to Firmicutes ratio between children with ASD and typically developing children. The tertiary outcome will be the difference in the diet quality in terms of lower dietary index, lower dietary diversity score and lower intake of fibre, iron, calcium, zinc and vitamin C in children with ASD and typically developing children.

ELIGIBILITY:
Inclusion Criteria for Cases:

Families with their children diagnosed with ASD by paediatrician or clinical psychologist according to the standard of the fourth or fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV or DSM-V) will be included.

Exclusion Criteria for Cases:

Families will be excluded if their children have the following conditions.

* Diagnosed with chronic seizures
* Suffered from recent infection 1-month prior to data and sample collection
* With diseases or disorders that affect dietary/physical activity habits (e.g. diabetes, cystic fibrosis, cerebral palsy)
* Usage of antibiotics and antifungal medications 1-month prior to data and sample collection
* Currently participating or have recently participated (i.e. 1-month prior to data and sample collection) in any trials or dietary intervention programs
* With other major medical or psychological illness, as judged by the investigators as ineligible to participate

Inclusion Criteria for Controls:

Families with typically developing children matched by child's age (i.e. within 6 months of age) and sex will be included. Children without ASD, delays in motor and language development, as well as behaviors as reported by their parents, and those do not have first-degree relatives with ASD will be included. Parents will also be asked to complete the Chinese validated version of Social Responsiveness Scale (SRS). For children who are screened with positive results, they will be further assessed by a developmental pediatrician to ascertain the autistic status. Only those who are screened negative, or those who are screened positive but subsequently ascertained by the developmental pediatrician being free from autistic symptoms will be included.

Exclusion Criteria for Controls:

The exclusion criteria will be same as those for the families with children of ASD.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Sixty five families with children of ASD of Chinese origin aged between 3 and 6 years and 65 control families with typically developing children matched by child's age (within 6 months) and sex will be recruited through invitation letters using a convenience sampling method in nurseries and kindergartens, in particular those with integrated programmes for ASD children. Some other possible channels for recruiting families with ASD children will include non-governmental organizations (NGOs) and some ASD family supporting groups.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2017-11-04 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Mealtime behaviours | baseline
  Mealtime behaviours measured using the Chinese version of the Brief Autism Mealtime Behaviour Inventory

SECONDARY OUTCOMES:
Gastrointestinal symptoms | baseline
  Gastrointestinal symptoms measured using the Chinese version of the Questionnaire on Pediatric Gastrointestinal Symptoms - Rome III (QPGS-RIII)
Gut microbiota profile | baseline
  Gut microbiota profile measured using 16s sequencing

OTHER OUTCOMES:
Current diet quality | baseline
  Current diet quality measured using 3-day diet record
Usual diet quality | baseline
  Usual diet quality measured using food frequency questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, China